CLINICAL TRIAL: NCT04812743
Title: Colorectal Health Research Champions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of grant funding
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19-15899; HM20017398 (Other: Virginia Commonwealth University IRB); NCI-2019-08595 (Other: NCI)
Record Dates: First submitted 2020-12-16; First posted 2021-03-24 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Colon; Cancer of Rectum
Keywords: Prevention
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal Health Research Champion trainees (Experimental): Colorectal Health Research Champion (CHRC) trainees receive 5 education sessions on colorectal cancer, clinical research, biospecimen donation, ethics, and presentation skills. The CHRCs will invite others in their social networks to present to them this educational information, following the train the trainer model of health education.
  Interventions: Behavioral: Colorectal Health Research Champions

INTERVENTIONS:
Behavioral: Colorectal Health Research Champions — 20 Colorectal Health Research Champions will be recruited from the VCU Massey Cancer Center Catchment Area (66 counties in Virginia) The Colorectal Health Research Champions will receive training in four specific areas during group educational sessions.
  Colorectal Health Research Champions will be asked to disseminate the four defined messages on at least two occasions to small groups in their social network in a venue of their choice (house chats, faith-based, social gatherings, family gatherings, etc.). We ask that each CHRC participant host 2 chats with 5-10 people in attendance at each chat. We expect that at least 200 participants will be invited to chats through 10 CHRCs.

SUMMARY:
The purpose of the Colorectal Health Research Champions program is to provide accurate and reliable colorectal health cancer information that they can share within their communities to encourage cancer prevention, screening, and early detection, as well as the importance of participating in research.

ELIGIBILITY:
Inclusion Criteria:

the individual is > 30 years of age

* They are literate
* They are/were directly or indirectly impacted by colorectal cancer and interested in becoming a champion for colorectal cancer research.

To participate in a chat hosted by the CHRC the inclusion criteria is:

* adult of any gender
* over 30 years of age.

Exclusion Criteria for chat hosted by the CHRC:

-Those < 30 years of age

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Increase in participants knowledge and intentions related to colorectal cancer screening. | 4 months
  Participant knowledge will be measured using pre/post questionnaires, with each correct answer being worth one point (14 total points) Higher summary scores indicate a greater change in knowledge. Intentions are measured on a 5 -point likert scale.
Increase in knowledge and intentions related to biospecimen donation and clinical trial participation. | 4 months
  Participant knowledge and intentions related to biospecimen donation and clinical trial participation will be measured using pre/post questionnaires, with each correct answer being worth one point (20 total points). Higher summary scores indicate a greater change in knowledge. Intentions are measured on a 5 -point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa B Sheppard, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT04812743/ICF_000.pdf